CLINICAL TRIAL: NCT02506075
Title: Effectiveness of Transcranial Direct Current Stimulation for Unilateral Neglect After Stroke
Brief Title: A Study of tDCS for Unilateral Neglect in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University (Other)
Collaborators: Medwill hospital (Unknown)
Responsible Party: Principal Investigator, Yong-il Shin, Associate Professor, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNUYH-03-2015-005
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-tDCS group (Experimental): In Pre-tDCS group, total sessions of the transcranical direct current stimulator stimulation(tDCS) was done for each three subgroups and visual inattention training was followed after that.
  Patient had 2 times of tDCS for 13 minutes with 20minutes of resting interval. After that, additional 2 times of Visual inattention training was done with same protocol.
  Interventions: Device: Transcranical direct current stimulator; Behavioral: Visual inattention training
- Simultaneous tDCS group (Experimental): In Simultaneous transcranical direct current stimulator(tDCS) group, tDCS and visual inattention training was done simultaneously.
  Interventions: Device: Transcranical direct current stimulator; Behavioral: Visual inattention training
- Sham control group (No Intervention): without transcranical direct current stimulator(tDCS) or without visual training

INTERVENTIONS:
Device: Transcranical direct current stimulator — approved by Conformity European as safe treatment device for stroke patients
  Arms: Pre-tDCS group; Simultaneous tDCS group
Behavioral: Visual inattention training
  Arms: Pre-tDCS group; Simultaneous tDCS group

SUMMARY:
The primary objective of this study is to confirm and compare the effect of methods of transcranial direct current stimulation(tDCS) in the unilateral neglect of stroke patients

DETAILED DESCRIPTION:
Total 105 patients were recruited and randomized to receive either real or sham-tDCS. Real experimental groups were divided into two types; Pre-tDCS group and Simultaneous tDCS group. Two groups are again divided into three groups; Dual stimulation group, Unilateral stimulation group and Sham control group, respectively.

In Pre-tDCS group, total a sessions of the tDCS stimulation was done for each three subgroups and visual inattention training was followed after that. In Simultaneous tDCS group, tDCS and visual inattention training was done simultaneously. For each subgroups, tDCS was attached at following locations; unilateral cathodal tDCS on unaffected PPC(postparietal cortex), P3 , dual cathodal tDCS on P3 and anodal tDCS on affected PPC, P4.

The patients were initially evaluated at baseline, immediately, 60min, 120min, 24 hrs after the training session.

ELIGIBILITY:
Inclusion Criteria

* Subjects who have diagnosed as primary stroke by physician's physical exam or radiologic diagnosis
* Subjects who have cortical or subcortical brain lesion
* Subjects ages older than 18years old
* Subjects who have 19 of K-MMSE score
* Subjects who has unilateral neglect with BIT-C less than 129
* Subjects who understand the purpose of the study and acquired the consent of the patient or caregiver
* Subjects who had no effect from brain stimulation or electrical stimulation therapy
* Subjects whose dominant side are confirm by Edinburgh Handedness Inventory

Exclusion criteria

* Subjects who have pre-existing and active major neurological disease
* Subjects who have pre-existing and active major psychiatric disease, such as major depression, schizophrenia, bipolar disease, or dementia
* Subjects who have brain lesion except cortex or subcortex area
* Subjects who have any metal component after brain surgery, low threshold to pain, history of seizure
* Subjects who is estimated as not appropriate for the study by the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Behavioral Inattention Test | up to 2 min
  Line bisection test
Behavioral Inattention Test | up to 2 min
  Letter cancellation test

SECONDARY OUTCOMES:
Behavioral Inattention Test | 60 min, 120 min, 24 hrs after intervention
  Line bisection test
Behavioral Inattention Test | 60 min, 120 min, 24 hrs after intervention
  Letter cancellation test
ADL assssement | 60 min, 120 min, 24 hrs after intervention
  Catherine Bergego Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Il Shin, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

REFERENCES:
- [Background] Adkins-Muir DL, Jones TA. Cortical electrical stimulation combined with rehabilitative training: enhanced functional recovery and dendritic plasticity following focal cortical ischemia in rats. Neurol Res. 2003 Dec;25(8):780-8. doi: 10.1179/016164103771953853. PMID 14669519